CLINICAL TRIAL: NCT01104129
Title: Detection of Pancreatic Cancer and Pre-cancer by Stool DNA Testing: A Feasibility Study
Brief Title: Stool Testing for Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: AAAD8007
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Intraductal Papillary Mucinous Neoplasm (IPMN); Stool-based digital melt curve (DMC) assay; Surgical resection for pancreatic cancer; Hereditary Pancreatic Cancer Syndrome; Genetic mutations linked to pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Dyggve-Melchior-Clausen syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tissue Collection: Fresh frozen resected tumor and IPMN tissue will be obtained whenever possible. All resected specimens, cancer and IPMN, will have histologic review to confirm the diagnosis. Ten slices of 10 microns each from each specimen will be prepared and sent to Mayo Clinic on dry ice.
  * Stool Collection: Prior to any surgery, stool will be collected from both study and control patients. Collection containers and mailing materials will be provided to subjects at time of their recruitment. Stool specimens will be mailed directly to Mayo Clinic within 48 hours of collection. Stool will be stored at 80 °C until assayed.
  * Stool DNA extraction: After stool is homogenized, crude stool DNA will be extracted and purified.
  * Digital melt curve mutation analysis: Target gene copies in captured stool DNA and tissue DNA will be quantified with real-time PCR. To target the mutations detected in tumor specimens, we will utilize PCR primers that scan for specific gene abnormalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Individual who has not had pancreatic cancer/IPMN; surgical resection for lesion of pancreas; history of colorectal, gastric cancer, esophageal, or head-and-neck cancer; administration of chemotherapy less than 1 week prior to enrollment; or an endoscopic procedure conducted less than 1 week prior to enrollment.
- Diagnosis of Pancreatic Cancer/IPMN: Patients diagnosed with Pancreatic Cancer/Intraductal Papillary Mucinous Neoplasm who are scheduled for surgical resection.

SUMMARY:
The purpose of this study is to determine if pancreatic cancer/pre-cancer can be detected in early stages through the molecular analysis of stool samples. Investigators hypothesize that analysis of stool samples using digital melt curve (DMC) analysis, can be used as a sensitive and specific method to detect the common genetic abnormalities present in pancreatic cancers and pre-cancerous lesions of the pancreas.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDC) remains the fourth leading cause of cancer-related death in the United States. This is largely due to the fact that most patients present with advanced, unresectable disease, highlighting the critical need for a screening test for this disease. Stool testing is an approach that has not been explored for use in PDC screening. With the advent of stool-based DNA tests, it may be possible to target genetic abnormalities that have been recently characterized in PDC tumorigenesis.

Aim: The aim of this study is to determine if deoxyribonucleic acid (DNA) alterations present in pancreatic cancer and precancerous intrapapillary mucinous neoplasms (IPMN) can be reliably recovered in matched stool.

Methods: This is a case-control prospective study to determine the utility of a stool-based digital melt curve (DMC) assay in PDC screening. A total of 30 patients (18 with pancreatic cancer, 12 with IPMN) who will be undergoing pancreatic resection will be enrolled. Pancreatic neoplastic tissue will be isolated from their surgical specimens and the genes most commonly mutated in PDC will be sequenced from extracted DNA. In addition, hypermethylation at common promoter sites will be assessed by methylation-specific PCR. The genetic and epigenetic alterations isolated in pancreatic tissue will be utilized as the targets for stool DMC assay. Blinded technicians will process stool specimens from control patients as well as a matched control. The primary outcomes of this study will be the sensitivity and specificity of the stool DMC assay in detecting genetic mutations present in tumor or IPMN lesions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Tissue-confirmed or radiological evidence of either pancreatic adenocarcinoma or intrapapillary mucinous neoplasm(IPMN).
* Scheduled for surgical resection of the adenocarcinoma or IPMN.
* Able to give informed consent

Exclusion Criteria:

* History of colorectal, gastric cancer, esophageal, or head-and-neck cancer.
* Endoscopic procedure conducted less than 1 week prior to enrollment.
* Unwillingness or inability to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with a diagnosis of pancreatic cancer/IPMN who are scheduled for surgical resection at Columbia University Medical Center's Pancreas Center will be accrued to this study.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Positive mutation rate in tumors/IPMN lesions vs. control | 30 days
  The positive mutation rates in tumor or IPMN lesions and in matched controls will be assessed.

SECONDARY OUTCOMES:
Percentage of patients with genetic abnormalities correctly detected in stool samples | 30 days
  Whether or not the genetic abnormalities that are detected in resected tissue can also be detected in stool specimens will be studied. If the hypothesis proves to be true, a new, non-invasive technique used in the detection of pre-cancerous lesions of the pancreas and pancreatic cancer will thereby be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K Chung, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No